CLINICAL TRIAL: NCT05068570
Title: The Effects of Arm Ergometry Training on Pulmonary Function in Children With Down Syndrome
Brief Title: Effect of Arm Ergometry on Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, hanaa mohsen, lecturer in the deparment of pediatrics and peditaric surgery , faculty of phyical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HANAA 8
Record Dates: First submitted 2021-09-07; First posted 2021-10-06 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: EFFECT OF ARM ERGOMETRY ON RESPIRATION

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERMINTAL GROUP (Experimental): start with cycle at a pace of 15-25 cycles per minute without resistance and end with cycle 45cycles per minute
  Interventions: Other: ARMEROMTERY
- CONTROL GROUP (No Intervention): selected respiratory exercise program

INTERVENTIONS:
Other: ARMEROMTERY — ARMERGOMTERY TRAINING FOR UPPERLIMB
  Arms: EXPERMINTAL GROUP

SUMMARY:
Cardiopulmonary issues are the major cause of sickness and hospitalisation in children with Down syndrome . Down syndrome children are also more likely to develop chronic lung infections, middle ear infections, and persistent tonsillitis.

DETAILED DESCRIPTION:
30 Down's syndrome children (boys and girls). randomly separated into two groups of equal size. Both groups received traditional chest physical therapy, with the addition of arm ergometry training in Group B

ELIGIBILITY:
Inclusion Criteria:

* comprehend and follow directions
* AGE 10-14

Exclusion Criteria:

Anomalies of the vasculature.

-Participating in sports of any kind. Moderate to severe asthma

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Discovery Spirometer | pre and post treatment for 14 weeks at 3 times per week.
  measure forced expiratory volume, the means incresed mean improvement
Discovery spirometer | Pre and post treatment for 14 weeks at 3 times per week
  Measure peak volume,the means incresed mean improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No